CLINICAL TRIAL: NCT01347853
Title: A Phase 3, Double-blind, Randomized Study of the Safety, Tolerability, and Analgesic Efficacy of Multiple Doses of Ketorolac Tromethamine Administered Intranasally for Postoperative Pain
Brief Title: Safety and Efficacy of Multiple Doses of Ketorolac Tromethamine Administered Intranasally for Postoperative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: David Bregman, M.D., Ph.D., Luitpold Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROX 2003-01
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac tromethamine (Experimental)
  Interventions: Drug: Ketorolac tromethamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac tromethamine — 30 mg intranasal post-surgery for up to 5 days total
  Arms: Ketorolac tromethamine
Drug: Placebo — Intranasal post-surgery for up to 5 days total
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled study in subjects who underwent major surgery. Each subject's study participation consisted of a screening visit and a treatment period of up to 5 days. Following surgery (Day 0), subjects were randomly assigned to receive intranasal ketorolac 30 mg or intranasal placebo when the pain intensity (PI) rating equaled at least 40 mm on a 100-mm visual analog scale (VAS). Subjects received study drug every 8 hours for 48 hours and then 3 times daily for up to 5 calendar days in total; the frequency of dosing could be reduced after 48 hours. Starting at the time of the first dose of study drug and continuing for the first 48 hours after surgery, the subjects had access to morphine sulfate (MS) administered via patient controlled analgesia (PCA). After PCA was no longer required, backup pain relief was provided by another standard nonsteroidal anti-inflammatory drug (non-NSAID) analgesic regimen. If the subjects were discharged before postoperative Day 4, they could self-medicate at home through postoperative Day 4. A safety follow-up evaluation was conducted by telephone approximately 14 days after the end of dosing in a subset of subjects (n = 60).

The primary objective was to evaluate the analgesic efficacy of multiple intranasal doses of ketorolac administered for up to 5 days. The secondary objective was to evaluate the safety and tolerability of this dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 years or older.
* Body weight > or = to 100 pounds and < or = to 300 pounds.
* Women of childbearing potential must have a negative serum pregnancy test result.
* Able to provide written informed consent.
* At least moderate pain as determined by a PI score of > or = to 40 mm on a 100-mm VAS.
* Expected to remain in the hospital for at least 48 hours with the possibility of remaining for 5 days.
* Willing and able to comply with all testing and requirements defined in the protocol.
* Willing and able to complete the post-treatment visit.

Exclusion Criteria:

* Allergy or sensitivity to ketorolac or EDTA.
* Allergic reaction to aspirin or other NSAIDs.
* Current upper respiratory tract infection or other respiratory tract condition that could interfere with the absorption of the nasal spray or with the assessment of adverse events.
* Use of any intranasal (IN) product within 24 hours prior to study entry.
* Clinically significant abnormality on screening laboratory tests.
* History of cocaine use resulting in nasal mucosal damage.
* Active peptic ulcer disease, recent (defined as within 6 months) history of peptic ulcer disease or gastrointestinal bleeding considered by the investigator to be clinically significant.
* Advanced renal impairment (serum creatinine > 1.5 mg/dL) or a risk for renal failure due to volume depletion.
* A history of any other clinically significant medical problem, which in the opinion of the investigator would interfere with study participation.
* Participation within 30 days of study entry or within 5 times the half- life, whichever is longer, in another investigational drug study.
* Allergy or significant reaction to opioids.
* Pregnancy or breastfeeding.
* Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-06; Primary Completion 2005-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The Summed Pain Intensity Difference (SPID) on Day 1 | 6 hours after drug administration
  Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. The PI values were obtained every hour following the first dose of study medication on Day 1. Pain intensity difference (PID) was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication. A summed PID (SPID) on the first postoperative day was calculated at 6 hours.

SECONDARY OUTCOMES:
Morphine sulfate consumption at 24 hours and 48 hours | 24 hours and 48 hours after drug administration
Hourly Pain Intensity Difference (PID) scores. | Hourly following the first dose of study medication up to 8 hours
  Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. The PI values were obtained during the first 8 hours following the first dose of study medication on Day 1. PID was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication.
Quality of analgesia | First dose of study medication on Day 1 to the first dose of MS by PCA
  Quality of analgesia was assessed on a 5-point categorical scale with 0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent.
Global assessment of pain control | 8 hours following first dose of study medication
  A global evaluation of pain control was conducted once daily at bedtime using a 5-point categorical scale on which 0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent.
Onset and duration of pain relief | 8 hours following first dose of study medication
  The onset of pain relief was defined as the time when the stopwatch was stopped to indicate "meaningful" pain relief. Peak PID was calculated. Duration of analgesia was defined as the time from the first dose of study medication on Day 1 to the first dose of MS by PCA.

CONTACTS AND LOCATIONS:
Locations (1):
- Waikato Clinical Research, Hamilton, New Zealand